CLINICAL TRIAL: NCT06240936
Title: Effects of Active Cycle of Breathing Techniques With and Without Acapella in COPD Patients
Brief Title: Active Cycle of Breathing Techniques With and Without Acapella in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0339
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; ACBTs; Acapella,; breathlessness; fatigue
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Active Comparator): ACBTs will be applied on the patients. It consist of the following three phases, breathing control,tboracic expension and forced expiration technique.
  Interventions: Other: Active Cycle of breathing
- Active Cycle of breathing with Acapela (Experimental): ACBTs will be applied on the patients. It consist of the following three phases, breathing control,tboracic expension and forced expiration technique. The Acapella device is a handheld device used to help loosen mucus in the lungs. Sit up straight and hold the device in the upright position. Take a deep breath in and seal lips around the mouthpiece. Exhaleforcefully through the mouthpiece, using your stomach muscles to push the air out. Repeat this process several times, taking breaks. After using Acapella cough to clear any mucus that has been loosened. Clean the device after each use.
  Interventions: Other: Active Cycle of breathing; Other: Active Cycle of breathing with Acapella

INTERVENTIONS:
Other: Active Cycle of breathing — Active Cycle of Breathing Techniques will be given to group A. In Active cycle of breathing exercises, breathing control, thoracic expansion and forced expiration technique will be applied. 3-4 sets of exercise ,10-15 mint, 4 times per week for 4 weeks.
Other: Active Cycle of breathing with Acapella — Acapella device will be used along active cycle of breathing techniques to group B. 3-4 sets ,10 mints foe acapella training ,15 -20 munts ,4 times per week for 4 weeks.
  This technique is active form of therapy in which patient uses its own energy on request to aid in treatment.
  Arms: Active Cycle of breathing with Acapela

SUMMARY:
Chronic Obstructive Pulmonary Disease refers to a group of progressive lung diseases the block air flow and make it difficult to breath. It is potentially fatal and fourth leading cause of death in the world. The symptoms of this condition include shortness of breath, frequent coughing, fatigued and tightness in the chest. Due to the secretions in the lungs sometime patients will have great difficulty catching the breath after walking or exercise. Patient will also feel breathless just sitting or relaxing. Active Cycle of breathing technique can be used to mobilize and clear secretions. It will improve their stamina and reduce the episodes of breathlessness, help to remove the secretions from the lungs and feel better overall. Acapella is a small hand held device which help to loosen and clear secretions from the chest it has both resistive and vibratory features. A randomized control trial will be conducted at Gosha e Shifa hospital and General hospital Lahore through convenience sampling technique on 42 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. Group A will be treated with active cycle of breathing exercises/techniques and Group B will be treated with Acapella device with active cycle of breathing exercise .Outcome measure will be conducted through Modified dyspnea scale, acapella device usage and questionnaire after 4 weeks and also perform Pulmonary function test .Data will be analyzed using SPSS software version 21. After assessing normality of data by Shapiro - wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups. Acapella device uses and active cycle of breathing technique will be applied for comparing their effect in patients of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women age between 35-50 years.
* Having smoking history .(1)
* Dyspnea MRC scale grade 2 and grade 3.(20)
* Gold standard COPD grade 2

Exclusion Criteria:

* Any kind of infective pulmonary condition .
* Restrictive lung disease.(20)
* Pregnancy.
* Any severe heart disease

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Modified Dyspnea scale. | baseline and fourth week
  Data collection tool for shortness of breath is modified dyspnea scale there will be 10 readings. It also accesses breathing discomfort, sensory qualities and emotional distress.
PFTs | baseline and fourth week
  The test will measure the lung volume, and ABGs. It is important tool for the investigation and monitoring of patients with respiratory pathology
Sputum diary BCSS | baseline and fourth week
  In this diary we will check breathlessness, cough and sputum. It also includes the score of patient wellbeing and documented all minor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Younis, MSPT (CP), Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anto JM, Vermeire P, Vestbo J, Sunyer J. Epidemiology of chronic obstructive pulmonary disease. Eur Respir J. 2001 May;17(5):982-94. doi: 10.1183/09031936.01.17509820. PMID 11488336
- [Background] Vogelmeier CF, Roman-Rodriguez M, Singh D, Han MK, Rodriguez-Roisin R, Ferguson GT. Goals of COPD treatment: Focus on symptoms and exacerbations. Respir Med. 2020 May;166:105938. doi: 10.1016/j.rmed.2020.105938. Epub 2020 Mar 21. PMID 32250871
- [Background] Lange P, Ahmed E, Lahmar ZM, Martinez FJ, Bourdin A. Natural history and mechanisms of COPD. Respirology. 2021 Apr;26(4):298-321. doi: 10.1111/resp.14007. Epub 2021 Jan 28. PMID 33506971